CLINICAL TRIAL: NCT06519214
Title: Correlation of Social Media Usage With Physical Activity and Academic Performance in School Aged Children
Brief Title: Correlation of Social Media Usage With Physical Activity and Academic Performance in Children
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/RCR&AHS/23/0784
Record Dates: First submitted 2024-06-11; First posted 2024-07-25 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Social Media Addiction
Keywords: social media; physical activity; academic performance; school
MeSH Terms: conditions — Internet Addiction Disorder; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Social media are internet-based applications that allow users to exchange messages or user-generated content for the purposes of social connection, entertainment, or education. WhatsApp, Skype, Facebook, Instagram, Telegram, and Twitter are a few of the most well-known and frequently used virtual social networks. In young children and school-age populations have concentrated on the correlation between watching television and playing video games and academic achievement, demonstrating a detrimental impact on physical health. Children who watch television for more than two hours a day tend to perform worse academically and engage in less physical activity.

DETAILED DESCRIPTION:
The study will be conducted as a non-probability convenience sampling with the objective of Social Media Usage on Physical Activity and Academic Performance in Young School-Age Individuals. Patient age range from 10 to 16 years, both genders.

Sample size is 289 students of private and government schools. Collaborate with schools within the selected age range and obtain permission for the study. The patients' assessment includes the use social media addiction scale, Academic performance questionnaire, SAMU DIS-FIT Battery. Data will be analyzed by SPSS version 26. Descriptive statistics will be checked by using frequency, percentage, mean and standard deviation of the variables. Normality of the collected data will be checked by using SPSS version 26. If p value will be more that 0.05 will apply parametric test. if it is less than 0.05 will apply non parametric test. Pearson correlation "r will be applied for parametric data and Spearmon RAO will be used for non-parametric data

ELIGIBILITY:
Inclusion Criteria:• Age of the participant will be 10 to 16 years.(3)

* Male and female both will be included.(25)
* Constantly using screen time with minimum 40 minutes per day.(5)
* Healthy and physical fit participant will be included. • Regular and enrolled students of public and private schools

Exclusion Criteria:

Children with disabilities that are limited in their ability to understand the instructions or the performance of the activities (Cognitive impairment etc.)

* Students with any significant past medical history or surgical history will not be included in this study

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: physical activity and academic performance with the sample size of 289 students of schools under age 10-16 years
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Academic performance questionnaire | 8 weeks
  measure academic performance of a child

SECONDARY OUTCOMES:
Bergen social media questionnaire | 8 weeks
  measure social participation of a child

CONTACTS AND LOCATIONS:
Overall Officials: Iqra Ali, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ceylan A, Demirdel E. The Relationship Between Academic Performance and Physical Activity, Smart Phone Use and Sleep Quality in University Students. Clinical and Experimental Health Sciences. 2023;13(3):549-54
- [Background] Martin JT, Acampad EM, Baligad RA, Larce A, Santos M, editors. Correlation of physical activity and social media use of students. Proceedings of the 2nd International Conference on Sports Science, Health and Physical Education; SCITEPRESS-Science and Technology Publications, Bandung, Indonesia; 2017.